CLINICAL TRIAL: NCT00794027
Title: The Clinical Outcomes Associated With a Modified Yoga Program in Heart Failure
Brief Title: The Effects of a Yoga Program in Heart Failure Patients
Acronym: YOGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H40997-33062-01
Record Dates: First submitted 2008-11-11; First posted 2008-11-19 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: heart failure; yoga; quality of life
MeSH Terms: conditions — Heart Failure | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga group (Other): Patients with heart failure
  Interventions: Behavioral: Yoga Classes

INTERVENTIONS:
Behavioral: Yoga Classes — 8 weeks of yoga training that occurs 2 times per week. The patients will also perform yoga breathing at home 3 times per week.
  Other Names: breathing
Behavioral: Yoga classes — Heart failure patients will undergo 8 weeks of yoga training 2 times per week and perform yoga breathing at home 3 times per week
  Other Names: pranyama

SUMMARY:
The proposed research will investigate the clinical outcomes associated with a modified yoga training program in patients with heart failure (HF). HF patients (15-20) will participate in a modified yoga program during an 8 week period, two times per week with instruction for home practice. Baseline measures and follow-up will be taken after 8 weeks. The underlying hypothesis to be tested is that yoga-induced improvements in nervous system and skeletal muscle function will yield positive effects on clinical outcomes, functional ability, and health-related quality of life in patients with HF.

The effect of combined yoga and breathing training on the natural history of HF and its potential to decrease negative clinical outcomes and improve symptoms is unknown. The relevance of this research is related to the important information it will provide to clinicians caring for patients with HF and will be the basis for pilot data for future NIH funding applications.

DETAILED DESCRIPTION:
The proposed research project is a pilot study designed to delineate the clinical outcomes associated with a modified yoga program in a population of adults with ventricular dysfunction and clinical heart failure (HF). The researchers hypothesize that patients in a modified yoga training program will have a significant improvement in clinical outcomes, functional ability, and health-related quality of life (HRQOL). The researchers propose to evaluate 15-20 subjects with chronic HF and New York Heart Association Functional Class (NYHA) II-III and obtain baseline physiological, functional, and HRQOL measurements. After obtaining baseline measurements, patients will participate in a modified yoga program with instruction for home practice for 8 weeks. Baseline measurements include: Vital signs, oxygen saturation, heart rate variability, exercise distance, muscular strength and flexibility determination, and various indices of HRQOL. At the conclusion of 8 weeks of yoga training the same measurements will be obtained.

In a group of chronic HF patients, the specific aims are the following:

1. To develop a safe and feasible yoga program;
2. To determine whether clinical outcomes (vital signs, oxygen saturation, heart rate variability), functional ability (exercise distance, muscular strength and flexibility determination), and HRQOL are positively affected by a modified yoga program.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class I-III
* normal sinus rhythm
* able to walk
* ability to read or understand English
* age 30-75

Exclusion Criteria:

* cognitive impairment
* inability to consent
* 100% paced with pacemaker
* hospitalization within 3 months
* MI or recurrent angina within 6 months
* severe stenotic valve disease
* history of sudden cardiac death
* history of uncontrolled ventricular tachyarrhythmias
* pulmonary hypertension
* FEV1 less than 1 liter by spirometry
* orthopedic impediments to yoga
* medication noncompliance

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Improvement in heart rate variability | 8 weeks

SECONDARY OUTCOMES:
Health-related quality of life | 8 weeks
muscle strength | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jill Howie-Esquivel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Osher Center and UCSF Cardiology Faculty Practice, San Francisco, California, United States